CLINICAL TRIAL: NCT06126965
Title: A Phase III, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of KX-826 for Topical Use in Chinese Adult Male Patients With Androgenetic Alopecia (AGA)
Brief Title: Phase III Study of KX-826 With Adult Male Patients With AGA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Collaborators: Suzhou Koshine Biomedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KX0826-CN-1003
Record Dates: First submitted 2023-10-29; First posted 2023-11-13 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-11

CONDITIONS: Androgenetic Alopecia
Keywords: KX-826; AGA
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KX-826-0.5% BID (Experimental): treatment dose group of 0.5% BID(0.5%)
  Interventions: Drug: KX-826-（5%） BID
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KX-826-（5%） BID — Dosage and administration: Topical application, 7 sprays (approximately 1 ml)/time, in the target area of the scalp, starting from the center of the affected area and massaging with hands until absorption. It should be used when the hair and scalp are completely dry. Wash hands after use. The randomized active drug would be administered to the scalp once in the morning and once in the evening.
  Other Names: KX-826-5 mg(5%)60mL BID
  Arms: KX-826-0.5% BID
Other: Placebo — Dosage and administration: Topical application, 7 sprays (approximately 1 ml)/time, in the target area of the scalp, starting from the center of the affected area and massaging with hands until absorption. It should be used when the hair and scalp are completely dry. Wash hands after use. The randomized matching placebo would be administered to the scalp once in the morning and once in the evening.
  Arms: Placebo

SUMMARY:
This is a phase III, multi-center, randomized, double-blind, placebo-controlled clinical study to evaluate the efficacy and safety of KX-826 for topical use in Chinese adult male patients with androgenetic alopecia (AGA).

DETAILED DESCRIPTION:
In this study, around 740 adult male subjects with AGA (rating IIIv, IV and V on Hamilton-Norwood scale) were to be enrolled. All subjects would be evaluated with 1:1 randomized to receive active drug or placebo in a double-blind fashion (370 subjects in each group), and would be treated for 24 weeks at the specified dose and frequency of each group. During the study, the subjects would undergo periodic efficacy and safety-related examinations and evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the study treatment regimen and visit plan, voluntarily enroll in the study, and sign the ICF in writing;
2. Male, ≥ 18 old;
3. Clinically diagnosed as androgenetic alopecia;
4. Rating IIIv, IV and V on Hamilton-Norwood scale;

Exclusion Criteria:

1. Have used androgen replacement therapy, immunosuppressants, corticosteroids and other drugs that may affect the efficacy evaluation within 3 months prior to screening;
2. Have used minoxidil within 6 months prior to screening;
3. Have used finasteride or dutasteride within 12 months prior to screening;
4. Had used topical drugs for alopecia sites within 3 months prior to screening;
5. Have received scalp radiation and/or laser or surgical therapy within 12 months prior to screening;
6. Those who, in the opinion of the investigator, have other conditions that may affect compliance or are not suitable for participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, aged ≥ 18 years, in good general health;
Enrollment: 740 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
change in non-vellus hair count in the target area (TAHC, mean change from baseline at Week 24 in comparison to placebo). | mean change from baseline after 24 weeks of treatment
  change in non-vellus hair count in the target area (TAHC, mean change from baseline at Week 24 in comparison to placebo).

SECONDARY OUTCOMES:
Secondary Outcome Measure: | change from baseline after 6, 12, 18, and 24 weeks of treatment, assessed using a 7-category method
  Hair growth assessment (HGA) of patient self-assessment, and Hair growth assessment (HGA) of investigator assessment
Change in non-vellus hair diameter (width) in the target area (TAHW) (change from baseline at Weeks 6, 12, 18, 24 of treatment) | change from baseline after 6, 12, 18, and 24 weeks of treatment
  Change in non-vellus hair diameter (width) in the target area (TAHW) (change from baseline at Weeks 6, 12, 18, 24 of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital; Qinping Yang, Principal Investigator — Huashan Hospital
Locations (26):
- China (26):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital,Cmu, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Sir Run Run Shaw Hospital,ZheJiang University School Of Medicine, Zhejiang, Hangzhou
  - The First Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Hospital Of Traditional Chinese And Western Medicine, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdou, Sichuan
  - Tianjin Academy Of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Affiliated Hangzhou First People's Hospital,Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang